CLINICAL TRIAL: NCT00628576
Title: Deep Venous Thrombosis. Long-Term Results After Treatment With Either Low-Molecular -Weight Heparin or Unfractionated Heparin. Examinations of the Venous System.
Brief Title: Evaluation of Long-Term Sequelae After Thrombophlebitis, i.e. Deep Venous Thrombosis of the Lower Extremities
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal investigator: Benedicte Laursen MD, DMSc, Department of Haematology and Medicine Aalborg Hospital, 9100 Aalborg, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VN 2003/15 (2-16-4 - 0001- 03)
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 2008-02

CONDITIONS: Deep Venous Thrombosis
Keywords: Deep Venous Thrombosis; lower extremities; Chronic Venous Insufficiency; Postthrombotic Syndrome; Heparins; Low-molecular- weight heparin; Tinzaparin
MeSH Terms: conditions — Venous Thrombosis; Postthrombotic Syndrome | interventions — Heparin; Tinzaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): UFH: patients treated with unfractionated heparin
  Interventions: Drug: unfractionated heparin
- 2 (Experimental): FH: patients treated with low-molecular-weight (fractionated) heparin
  Interventions: Drug: Tinzaparin (Leo)

INTERVENTIONS:
Drug: unfractionated heparin — UFH: Continuous i.v. infusion 100 IU/kg/4hrs initially and then adjusted to maintain APTT value 1.5 - 2.5 the pre-treatment value
  Other Names: Heparin SAD 1000 IU/ml
  Arms: 1
Drug: Tinzaparin (Leo) — FH (Tinzaparin): 175 iu/kg s.c. in the abdomen once daily
  Other Names: Innohep (Leo)
  Arms: 2

SUMMARY:
The purpose of the study was to evaluate efficacy and safety of the new acute treatment of deep venous thrombosis by use of low-molecular-weight heparin compared with standard treatment using unfractionated heparin, especially concerning long-term morbidity.

DETAILED DESCRIPTION:
Deep-venous thrombosis (DVT) remains a common clinical problem (annual incidence 0.10-0.16%) and long-term morbidity as chronic venous insufficience (CVI) in 10-30%.

As to recurrent DVT, initial treatment with Low-Molecular-Weight Heparin ( to-day's terminology Fractionated Heparin (FH)) and Unfractionated Heparin (UFH) has shown equal efficiency, whereas the efficacy concerning long-term morbidity has only more recently been published.

This study was initiated to compare the efficacy of UFH and FH concerning the incidence of CVI after symptomatic DVT at short-term and long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* First DVT with or without known risk factors except overt cancer
* Second DVT more than two years after the first if the patient was without clinical signs of CVI.

Exclusion Criteria:

* Contraindication to anticoagulation therapy
* Candidate to thrombectomy with arterious-venous fistula or thrombolytic therapy
* Known cancer at the time of the DVT diagnosis
* Patients unable to cooperate for anticoagulation therapy or manage the tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 1993-10; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of chronic venous insufficiency (CVI) - (Postthrombotic Syndrome) based on internationally accepted criteria. | Two years and 6 to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Benedicte Laursen, MD, DMSc, Principal Investigator — Department of Haematology; Aalborg Hospital, 9100 Aalborg, Denmark
Locations (1):
- Dept. of Haematology; Aalborg Hospital, Aalborg, North Denmark, Denmark